CLINICAL TRIAL: NCT04231058
Title: The Effects of Acu-TENS in the Non-pharmacological Treatment of Dyspnea in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Non-pharmacological Treatment of Dyspnea in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: COPD
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of sufficient staff to conduct the study
Sponsor: Azienda USL Toscana Nord Ovest (Other)
Collaborators: Auxilium Vitae Volterra (Other)
Responsible Party: Principal Investigator, Alessandro Tani, Doctor in Department of Anesthesia and Intensive Care Unit, Azienda USL Toscana Nord Ovest
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: USL area vasta NordOvest
Record Dates: First submitted 2019-12-16; First posted 2020-01-18 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Dyspnea
Keywords: COPD; Transcutaneous Electrical Nerve Stimulation
MeSH Terms: conditions — Dyspnea; Pulmonary Disease, Chronic Obstructive | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous Electrical Nerve Stimulation (TENS) (Experimental): 15 experimental subjects treated withTENS and Pulmonary Rehabilitation
  Interventions: Device: TENS and pulmonary rehabilitation
- Rehabilitation (No Intervention): 15 experimental subjects treated with Pulmonary Rehabilitation only

INTERVENTIONS:
Device: TENS and pulmonary rehabilitation — Three treatments with TENS per week for 3 weeks each , lasting 45 minutes
  Arms: Transcutaneous Electrical Nerve Stimulation (TENS)

SUMMARY:
Dyspnoea is one of the most important determinants of quality of life and often limits the activities of daily life, in subjects suffering from moderate-to-severe chronic obstructive pulmonary disease (COPD). Pharmachological treatment of dyspnoea is affected by several side effects and, in long-lasting treatments, a reduction of clinical efficacy may occur. Previous studies showed a reduction of perceived dyspnoea after trials of acupuncture or Transcutaneous Electrical Nerve Stimulation over acupoints (Acu-TENS).

In this study will be investigated the effect of Acu-TENS on lung function and dyspnoea in patients with moderate-to-severe COPD (Cronic Obstructive Pulmonary Disease).

DETAILED DESCRIPTION:
Aim of the study is to verify the effectiveness of treatment with Acu-TENS to reduce perceived dyspnoea in patients suffering from moderate-to severe COPD. Secondary aims are to investigate the effects of the above treatments on quality of life, exercise capacity, pulmonary lung function.

Thirty consecutive patients, admitted to Auxilium Vitae Rehabilitation Centre for intensive pulmonary rehabilitation (PR) programme, suffering from moderate-to-severe COPD, will be enrolled. Subjects will be randomly assigned to two groups with different treatments (n=15 group 1: experimental subjects - PR+Acu-TENS and n=15 group 2: control subjects - PR only) by sequential block randomization.

An intensive inpatient PR programme will be applied to all participants. The programme will include the optimisation of drug therapy and daily sessions of:

1. Supervised incremental exercises on a treadmill, a cycle,and an arm ergometer according to the protocol suggested by Maltais et al. until the achievement of 30 min of continuous exercise at an intensity that elicited dyspnoea at level 5 on a modified Borg scale starting from a workload corresponding to 50% of maximal workload achieved during an initial incremental test;
2. Abdominal, upper- and lower-limb muscle activities involving lifting of progressively increasing light weight and shoulder and full-arm circling;
3. Education;
4. Nutritional programs and psychosocial counselling, when appropriate. A multidisciplinary team of chest physicians, nurses, physical therapists, a dietician, and a psychologist offered care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate-to-severe COPD (ATS-ERS definition)
* Patients who have not participated in a respiratory rehabilitation program within the previous 3 months
* Patients admitted to the multi-specialist Rehabilitation Center Auxilium Vitae Volterra SPA for inpatient PR programme
* stable clinical conditions and absence of clinical deterioration, with stable dyspnea, cough and sputum; stability of blood gas values in the absence of signs of edema or heart failure
* Expression of informed consent valid for participation in the study
* Good collaboration in the activities foreseen by the study

Exclusion Criteria:

* Insufficient degree of cooperation
* Inability to walk independently
* Denial of informed consent to participate in the study
* patients with known serious cardiovascular diseases (unstable angina, advanced chronic heart failure, aortic aneurisms, etc.) contraindicating the inclusion in exercise training programmes; chronic neurological or musculoskeletal diseases impairing their ability to comply with study procedures; severe renal failure or end-stage dialysis, advanced cancer, epilepsy and other clinical conditions interfering with the procedures and the safety of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Baseline dyspnea evaluated with Baseline Dyspnea Index (BDI) | baseline
  Assessment of the perception of dyspnea with the basal dyspnea index (BDI) which measures the severity of dyspnea in a single state. The score ranges from 0 to 12. The lower the score, the worse the dyspnea severity
Transitional dyspnea evaluated with Transitional Dyspnea Index (TDI) | 2 week and 4 week
  Evaluation of the perception of dyspnea with a transitional dyspnea index (TDI) that measures changes in the severity of dyspnea compared to the baseline established by the Baseline Dyspnea Index (BDI). Rated from seven degrees ranging from -3 (major deterioration) to +3 (major improvement).

SECONDARY OUTCOMES:
Change in quality of life: SGRQ (St. George's Respiratory questionnaire) | baseline ,2 week and 4 week
  Change in quality of life evaluated with the SGRQ (St. George's Respiratory questionnaire)that is an instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Composed of 50 items .Total score ranging - 9 to + 9. The lower the score, the more deterioration in severichange inty of dyspnea
Change in functional capacity with the six-minute walk test (6mwt) | baseline , 2 and 4 week
  The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes .
Change in respiratory volumes | baseline, 2 and 4 week
  Variation of Forced expiratory volume in 1 second (FEV1), Forced vital capacity (FVC), Vital capacity (VC) and Forced expiratory volume in the 1st second (FEV1)
Change in respiratory muscle function | baseline, 2 and 4 week
  Variation of MIP (Maximal Inspiratory Pressure) and MEP (Maximal Expirator Pressure)
Change in lung diffusion capacity | baseline, 2 and 4 week
  Variation of Diffusing capacity (DLCO)
Impact of the disease | baseline, 2 and 4 week
  Impact of the disease will be evaluated by the CAT (Chronic Obstructive Pulmonary Disease Assessment Test).
  CAT are simple questionnaires that may be used to determine the severity of symptoms. Scores on CAT range from 0-40 with the higher the score, the more severe the disease
Patient's dissociative experience related to the stress measured with the Dissociative Experiences Scale (DES) | baseline, 2 and 4 week
  The Dissociative Experiences Scale (DES) is a psychological self-assessment questionnaire that measures dissociative symptoms. It contains twenty eight questions in which a percentage answer from 0 to 100% is given for each.
  The overall result, in percentage from 0 to 100, is obtained by dividing the sum of the percentage of each individual question by 28 which is the total number of questions.
  Patients with scores over 30 will be diagnosed with having dissociative identity disorder

CONTACTS AND LOCATIONS:
Overall Officials: Guido Vagheggini, MD, Principal Investigator — Azienda USL Toscana Nordovest, Fondazione Volterra Ricerche ONLUS
Locations (1):
- Santa Maria Maddalena Hospital, Volterra, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mazzoleni S, Montagnani G, Vagheggini G, Buono L, Moretti F, Dario P, Ambrosino N. Interactive videogame as rehabilitation tool of patients with chronic respiratory diseases: preliminary results of a feasibility study. Respir Med. 2014 Oct;108(10):1516-24. doi: 10.1016/j.rmed.2014.07.004. Epub 2014 Jul 16. PMID 25087837
- [Background] Celli BR, Decramer M, Wedzicha JA, Wilson KC, Agusti AA, Criner GJ, MacNee W, Make BJ, Rennard SI, Stockley RA, Vogelmeier C, Anzueto A, Au DH, Barnes PJ, Burgel PR, Calverley PM, Casanova C, Clini EM, Cooper CB, Coxson HO, Dusser DJ, Fabbri LM, Fahy B, Ferguson GT, Fisher A, Fletcher MJ, Hayot M, Hurst JR, Jones PW, Mahler DA, Maltais F, Mannino DM, Martinez FJ, Miravitlles M, Meek PM, Papi A, Rabe KF, Roche N, Sciurba FC, Sethi S, Siafakas N, Sin DD, Soriano JB, Stoller JK, Tashkin DP, Troosters T, Verleden GM, Verschakelen J, Vestbo J, Walsh JW, Washko GR, Wise RA, Wouters EF, ZuWallack RL; ATS/ERS Task Force for COPD Research. An official American Thoracic Society/European Respiratory Society statement: research questions in COPD. Eur Respir Rev. 2015 Jun;24(136):159-72. doi: 10.1183/16000617.00000315. PMID 26028628
- [Background] Montagnani G, Vagheggini G, Panait Vlad E, Berrighi D, Pantani L, Ambrosino N. Use of the Functional Independence Measure in people for whom weaning from mechanical ventilation is difficult. Phys Ther. 2011 Jul;91(7):1109-15. doi: 10.2522/ptj.20100369. Epub 2011 May 19. PMID 21596958
- [Background] Maltais F, LeBlanc P, Jobin J, Berube C, Bruneau J, Carrier L, Breton MJ, Falardeau G, Belleau R. Intensity of training and physiologic adaptation in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1997 Feb;155(2):555-61. doi: 10.1164/ajrccm.155.2.9032194.
- [Result] Ngai SP, Spencer LM, Jones AY, Alison JA. Acu-TENS Reduces Breathlessness during Exercise in People with Chronic Obstructive Pulmonary Disease. Evid Based Complement Alternat Med. 2017;2017:3649257. doi: 10.1155/2017/3649257. Epub 2017 Feb 20. PMID 28303156
- [Result] Ngai SP, Jones AY, Hui-Chan CW, Ko FW, Hui DS. Effect of 4 weeks of Acu-TENS on functional capacity and beta-endorphin level in subjects with chronic obstructive pulmonary disease: a randomized controlled trial. Respir Physiol Neurobiol. 2010 Aug 31;173(1):29-36. doi: 10.1016/j.resp.2010.06.005. Epub 2010 Jun 16. PMID 20601209
- [Result] Lau KS, Jones AY. A single session of Acu-TENS increases FEV1 and reduces dyspnoea in patients with chronic obstructive pulmonary disease: a randomised, placebo-controlled trial. Aust J Physiother. 2008;54(3):179-84. doi: 10.1016/s0004-9514(08)70024-2. PMID 18721121
- [Result] Yu M, Gao L, Kong Y, Yan Y, Shi Q, Si D, Bao H, Sun H, Li L, Li Y. Safety and efficacy of acupuncture for the treatment of chronic obstructive pulmonary disease: A systematic review protocol. Medicine (Baltimore). 2019 Sep;98(37):e17112. doi: 10.1097/MD.0000000000017112. PMID 31517846
- [Result] Suzuki M, Muro S, Ando Y, Omori T, Shiota T, Endo K, Sato S, Aihara K, Matsumoto M, Suzuki S, Itotani R, Ishitoko M, Hara Y, Takemura M, Ueda T, Kagioka H, Hirabayashi M, Fukui M, Mishima M. A randomized, placebo-controlled trial of acupuncture in patients with chronic obstructive pulmonary disease (COPD): the COPD-acupuncture trial (CAT). Arch Intern Med. 2012 Jun 11;172(11):878-86. doi: 10.1001/archinternmed.2012.1233. PMID 22905352